CLINICAL TRIAL: NCT06911710
Title: The Application of CAR-T Cell Therapy in Relapsed and Refractory Malignant Hematologic Tumors
Acronym: CAR-T
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Yihao Wang, chief physician, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2022-YX-013-01
Record Dates: First submitted 2025-03-23; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma, B-cell, Aggressive Non-Hodgkin (B-NHL); AML (Acute Myelogenous Leukemia); Myeloma Multiple; B-ALL; T-ALL/Lymphoma; T-lymphocyte Lymphoma
MeSH Terms: conditions — Lymphoma; Leukemia, Myeloid, Acute; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): CAR-T Cells infusion（CAR 2219，CAR2019，CAR19 ect）
  Interventions: Drug: CAR-T Cells infusion（CAR2219,CAR2019, CAR19 etc）

INTERVENTIONS:
Drug: CAR-T Cells infusion（CAR2219,CAR2019, CAR19 etc） — Phase I study: dose-escalation component.This part follows the "3+3" dose-escalation model, with 5 dose groups: 1×10^6, 1.5×10^6, 2×10^6, 2.5×10^6, 3×10^6 CAR+ cells/kg (different target CAR-T can be adjusted by the investigator according to the dose used in the previous clinical trial). Each dose group enrolled 3~6 patients with relapsed/refractory hematological diseases respectively, totaling 15~30 subjects, in order to evaluate the safety of CAR-T cells for the treatment of relapsed/refractory malignant hematological neoplasms and to determine the MTD. Phase II study: dose-expansion portion. After the MTD was confirmed, in the dose-expansion portion of the study (Phase II), it was expected that 65~60 subjects would receive the CAR-T cell injection infusion under RP2D to further evaluate the efficacy of CAR-T cell injection.

SUMMARY:
This study is an open, single-arm, prospective, Phase I/II clinical study using "3+3" dose escalation and dose expansion to investigate the safety, maximum tolerated dose, in vivo pharmacokinetic profile, and preliminary efficacy of CAR-T cell injections for the treatment of relapsed/refractory malignant hematological neoplasms in subjects.

ELIGIBILITY:
Inclusion Criteria:

With their own consent and have signed an informed consent form, willing and able to comply with the planned visits, study treatment, laboratory tests and other experimental procedures; Patients with recurrent/refractory malignant hematologic tumors as determined by clinical diagnosis; Age 18 years and above, both male and female; Subjects with a physical status of 0~2 on the Eastern Cooperative Oncology Group (ECOG) score; Expected survival >3 months from the date of informed consent; HGB ≥ 60g/L (transfusion is allowed); Liver and kidney function, cardiopulmonary function meet the following requirements: a) creatinine ≤1.5×ULN;b) Left ventricular ejection fraction ≥50%; c) Blood oxygen saturation >90%;d) Total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN; Subjects with pregnancy plans must agree to use contraception prior to enrollment in the study and after the study has lasted for six months; subjects should notify the investigator immediately if they become pregnant or suspect pregnancy.

Subjects in the different cohorts will still be required to fulfill the following conditions:

Lymphoma Cohort:

B-cell lymphoma Diagnosis of CD19+ and/or CD20+ and/or CD22+ and/or BAFF+ B-cell lymphoma confirmed by pathology and histology; Inert B-cell lymphoma (CLL, FL, MZL, LPL, HCL); Aggressive B-cell lymphoma (DLBCL, BL, MCL).

Meet the following criteria for relapsed or refractory B-cell lymphoma (meet 1 of the first 2 plus 3 below):

Less than 50% tumor shrinkage or disease progression after 4 courses of standard regimen regulated chemotherapy; relapse after achieving CR after standard regimen chemotherapy; subjects must have received adequate prior therapy, including at least: Anti-CD20 monoclonal antibody; Anthracycline-containing combination chemotherapy. T-cell lymphoma

Diagnosis of CD7+ refractory/relapsed T-lymphocyte lymphoma confirmed by pathology and histology, meeting any of the following criteria:

Relapsed: Disease relapse determined after having previously received at least two standardized treatment regimens to achieve complete remission, or disease relapse after having undergone stem cell transplantation to achieve complete remission; Refractory: previous treatment with at least two regimens and failure to achieve complete remission after the last treatment, or failure to achieve remission or disease progression after stem cell transplantation.

II Acute lymphoblastic leukemia cohort:

Acute B-lymphoblastic leukemia Refractory/relapsed B-lymphoblastic leukemia diagnosed as CD19+ and/or CD20+ and/or CD22+ and/or BAFF+ confirmed by immunohistochemistry or flow cytometry.

Refractory/relapsed B-lymphoblastic leukemia (meeting 1 of the following 4 criteria is sufficient):

Relapse within 6 months of first remission; first refractory without achieving complete remission with 2 cycles of standard chemotherapy regimen; failure to achieve complete remission or relapse after first or multiple lines of salvage chemotherapy; those who are not suitable for HSCT, or who have abandoned HSCT due to medical constraints, or those who have relapsed after HSCT.

Acute T-lymphoblastic leukemia

Diagnosis of CD7+ refractory/relapsed T-ALL/LBL confirmed by immunohistochemistry or flow cytometry, meeting any of the following criteria:

No CR after standard chemotherapy; CR after first treatment, but CR lasted less than 12 months; No CR after first or more remedial therapy; Relapse two or more times.

III. multiple myeloma cohort:

Positive expression of BCMA and/or CD19 and/or GPRC5D in myeloma cells by flow or immunohistochemistry; Patients with relapsed/refractory multiple myeloma who have received at least 1 prior therapy (including proteasome inhibitors (PIs) and immunomodulatory drugs (IMiDs)) or are resistant to proteasome inhibitors and/or immunomodulatory agents.

IV. myeloid tumor cohort:

Positive tumor cell antigen test results (CD7 and/or CD19 and/or CD47) confirmed by immunohistochemistry or flow cytometry; Diagnosis of myeloid tumors, including but not limited to AML and MDS, confirmed by pathology and the patient meets the following

Relapse or refractory requirements:

Relapse: reappearance of leukemic cells in the peripheral blood, or >5% of primitive cells found in the bone marrow, or extramedullary relapse after second-line or higher salvage therapy to achieve CR/CRi; Refractory: failure to achieve CR/CRi after at least 2 cycles of standard chemotherapy.

Exclusion Criteria:

a history of severe cardiac insufficiency with a left ventricular ejection fraction <50%; A history of severe lung function-impairing disease; Combination of other malignant tumors in progressive stages; Combination of severe infections that cannot be effectively controlled; Combination of severe autoimmune disease or congenital immunodeficiency; Active hepatitis (Hepatitis B virus deoxyribonucleic acid [HBV-DNA] or Hepatitis C virus ribonucleic acid [HCV-RNA] test results above the lower limit of detection); Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection; History of severe allergy to biological products (including antibiotics); Allogeneic hematopoietic stem cell transplantation patients who still have acute graft-versus-host reaction (GvHD) one month after stopping immunosuppressive drugs; Presence of other serious physical or mental illnesses or abnormal laboratory tests that may increase the risk of participation in the study or interfere with the results of the study, as well as patients who, in the opinion of the investigator, are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events | Day 28

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
Complete response rate (CRR) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
Duration of response (DOR) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
Progression free survival (PFS) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
Overall survival (OS) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up

OTHER OUTCOMES:
Kinetics of CAR-T cells | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
  Use flow cytometry or Q-PCR to monitor the kinetics of CAR-T cells.

CONTACTS AND LOCATIONS:
Locations (1):
- TianJin China. TianJin Medical University General, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No